CLINICAL TRIAL: NCT04800276
Title: Adapted Physical Activity in Patients With Lower Limb Peripheral Arterial Disease (ACTIV'AO)
Brief Title: Adapted Physical Activity in Patients With Lower Limb Peripheral Arterial Disease
Acronym: ACTIV'AO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHM-2019/S18/09
Record Dates: First submitted 2021-03-12; First posted 2021-03-16 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease, Adapted Physical Activity
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Two parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APA with consideration of ischemia localization (Experimental)
  Interventions: Other: muscle strengthening targeted on ischemic areas
- APA without consideration of ischemia localization (Experimental)
  Interventions: Other: global muscle strenghtening

INTERVENTIONS:
Other: muscle strengthening targeted on ischemic areas — muscle strengthening targeted on ischemic areas
  Arms: APA with consideration of ischemia localization
Other: global muscle strenghtening — global muscle strenghtening
  Arms: APA without consideration of ischemia localization

SUMMARY:
The prevalence of peripheral arterial disease is 12.2% in France. Intermittent claudication is the most common symtom of this disease. During physical exercise, such as walking, blood oxygen (O2) requirements increase. The development of atherosclerosis in the lower limbs, causes narrowing of the arteries and limits the increase in blood flow required for muscular effort. Patients then experience muscle pain, the intensity of which gradually increases until it forces them to stop. After stopping, the pain subsides and disappears in less than 10 minutes.

The location of the pain (calves and/or thighs and/or buttocks) is related to the location of the ischemia (distal in the calf, proximal in the thigh or buttock, or proximo-distal if several locations). This can have different consequences on the biomechanical parameters of walking and muscle activity. To date, the impact of this localization on physical capacity has never been studied.

These limitations are very disabling and impact the quality of life of patients.

In addition, poor lower limb performance is associated with higher mortality. Reducing symptomatology and improving functional abilities is therefore a major issue in patients with peripheral arterial disease. This can be achieved through the practice of an Adapted Physical Activity, an essential recommendation in the care of patients with peripheral arterial disease.

Our main hypothesis is that the physical activity rehabilitation protocol "Activ'AO" will improve the functional capacities of patients with peripheral arterial disease who have followed the program with the localization of ischemia with a greater consideration than in patients in the group following a "standard" APA protocol. Improvements in functional abilities (such as walking) will lead to improvements in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Lower Limb Peripheral Arterial Disease with IPSC < 0.90, arterial stenosis in the lower limbs and intermittent claudication
* No contraindication to physical activity

Exclusion Criteria:

* Severe or unstable cardiopulmonary pathologies, contraindicating exercise training
* Unstable angina or myocardial infarction <3 months
* Severe rheumatological pathology of the lower limbs
* Amputee of a lower or upper limb fitted with a device
* Extensive dermatosis of the lower limbs
* Known NYHA grade III or IV heart failure
* Known severe respiratory pathology
* Parkinson's disease, hemiplegia or paraplegia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Assess efficacity of Adapted Physical Activity with localization of ischemia on maximum walking distance compared to Adapted Physical activity without localization of ischemia | 12 weeks after inclusion
  The efficacity of Adapted Physical Activity was assessed by measure of maximum walking distance

SECONDARY OUTCOMES:
Assess efficacity of Adapted Physical Activity with localization of ischemia on walking abilities compared to Adapted Physical activity without localization of ischemia | 12 weeks after inclusion
  The efficacity of Adapted Physical Activity was assessed by measure of walking speed with actimeter
Assess efficacity of Adapted Physical Activity with localization of ischemia on static balance compared to Adapted Physical activity without localization of ischemia | 12 weeks after inclusion
  The efficacity of Adapted Physical Activity was assessed by measure of balance static with stabilometry Platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France